CLINICAL TRIAL: NCT06651437
Title: A Nutritional Questionnaire in an Adult Italian Hypertensive Population: Effects on Sodium and Potassium Intake (MINISAL-SIIA STUDY)
Brief Title: Salt Consumption After the Administration of Rapid Questionnaire (MINISAL-SIIA STUDY)
Acronym: MINISAL-SIIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Ferruccio Galletti (Other)
Responsible Party: Sponsor-Investigator, Prof. Ferruccio Galletti, Principal investigator, Federico II University
Organization: Federico II University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: FedericoIIEC/5516
Record Dates: First submitted 2024-09-05; First posted 2024-10-21 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): the Control group will not receive any additional information on diet
- Dietary educational intervention (Experimental): The dietary educational intervention group received dietary education to gradually reduce salt intake (a brief dietary education on the health damage due to excess salt consumption and on behavioural methods to gradually reduce dietary intake, for example at home, reduce the consumption of processed foods, do not bring salt shaker on the table, limit the use of condiments with a high sodium content; out of home, both when eating and when shopping, reduce the consumption of processed foods, check nutritional labels and choose products with lower salt content). In addition, written information was provided.
  Interventions: Other: Experimental dietary educational intervention

INTERVENTIONS:
Other: Experimental dietary educational intervention — At the end of the baseline examination, the Experimental group received a brief dietary education on the health damage due to excess salt consumption and on behavioural methods to gradually reduce dietary intake, for example at home, reduce the consumption of processed foods, do not bring salt shaker on the table, limit the use of condiments with a high sodium content; out of home, both when eating and when shopping, reduce the consumption of processed foods, check nutritional labels and choose products with lower salt content. In addition, written information was provided. All participants will be clinically followed every month, with potential titration of the antihypertensive therapy. After 3 months of follow-up, the baseline measurements will be carried out again. During the entire study period, subjects will be asked to maintain their lifestyle and report using additional medications.
  Other Names: Dietary educational intervention
  Arms: Dietary educational intervention

SUMMARY:
A strong and well-known association exists between salt consumption, potassium intake, and cardiovascular diseases. MINISAL-SIIA results showed high salt and low potassium consumption in Italian hypertensive patients. In addition, a recent Italian survey showed that the degree of knowledge and behavior about salt was directly interrelated, suggesting a key role of the educational approach. Therefore, the present study will aim to evaluate the efficacy of a short-time dietary educational intervention (MINIMAL-ADVICE) on sodium and potassium intake in hypertensive patients.

DETAILED DESCRIPTION:
High salt consumption is an important determinant of high blood pressure (BP) and cardiovascular diseases. Several intervention studies showed that a reduction in salt consumption reduces BP and can reduce cardiovascular risk beyond the beneficial effect on BP in people with and without hypertension. The World Health Organization (WHO) recommends that adults should consume no more than 5 g of salt daily. However, the mean daily intake of salt in the majority of countries worldwide exceeds this recommendation. In contrast to salt, epidemiological and intervention studies suggest beneficial effects of dietary potassium on BP and cardiovascular risk. This effect seems more pronounced during high salt consumption. The WHO currently also recommends that adults should consume not less than 90 mmol of potassium daily. However, also for potassium the WHO recommendations are not generally met.

Several countries have made some progress towards reducing habitual salt intake through a voluntary or regulatory approach, achieving a reduction of BP and cardiovascular disease in the young population. Our previous observational data detected that Italian general population samples consumed high dietary salt and low dietary potassium, far from the WHO guidelines recommendation. Excess dietary salt intake in the hypertensive patients' population was observed in all age categories and there were no differences in salt intake among different regions. Likewise, in the same hypertensive population the adequate potassium intake in both men and women, in all age categories, and in all the regions surveyed was much below the recommendation. These results point out the potential target to improve BP and cardiovascular risk, in particular in hypertensive patients. An Italian survey of a large cohort of the general population showed that the degree of knowledge and behaviour about salt was directly interrelated. These data suggested that educational approach is crucial to improve the level of salt consumption. The reduction of salt intake has been recommended by WHO as a cost-effective action that should be undertaken. Hence, an intervention study targeted to reduce dietary salt intake and also to increase dietary potassium consumption by an educational intervention is needed.

Given these premises, the aim of the present intervention study will be to evaluate the effect of a brief educational intervention "MINIMAL-ADVICE" for improving dietary salt and potassium intake in a hypertensive population. In addition, the effect of the educational intervention on BP in relation to the potential variation of salt and potassium intake will be also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adult hypertensive patients with essential hypertension
* assessment of organ damage
* and stable antihypertensive treatment (lifestyle modifications and/or drug therapy) for at least 6 months

Exclusion Criteria:

* patients with alteration in nutritional and absorptive status
* glomerular filtration rate lower than 60 ml/min/1.73 m2
* personal history positive for a recent cardiovascular event (less than 6 months)
* atrial fibrillation or flutter, frequent atrial or ventricular premature contractions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Urinary Sodium and Potassium excretion (mmol/24h) | 3 months
  Urinary sodium and potassium concentrations (mmol/24h) were measured by ion selective electrode potentiometry and urinary creatinine by a kinetic Jaffe reaction using an ABX Pentra 400 apparatus (HORIBA ABX, Rome, Italy). Quality control was effected using urine-specific reference samples from UrichemGol BIODEV (Milan, Italy).

SECONDARY OUTCOMES:
Systolic and Diastolic Blood Pressure (mmHg) | 3 months
  Systolic and diastolic BP were measured with automatic validated devices, after having the participant sit for at least 10 minutes. Three measurements of BP and heart rate were made at 2-minute intervals with the patient in the sitting position, and the average of the second and third readings was recorded. In addition, two measurements were made after 2 minutes in the standing position

REFERENCES:
- [Derived] D'Elia L, Strazzullo P, Del Giudice A, Desideri G, Di Quattro R, Ferri C, Grossi A, Malatino L, Mallamaci F, Maresca A, Meschi M, Casola A, Nazzaro P, Pappaccogli M, Rabbia F, Sala C, Galletti F; MINISAL-SIIA Study Group. "Minimal-Advice" on Salt Intake: Results of a Multicentre Pilot Randomised Controlled Trial on Hypertensive Patients. High Blood Press Cardiovasc Prev. 2025 Mar;32(2):181-190. doi: 10.1007/s40292-025-00704-1. Epub 2025 Jan 30. PMID 39883400